CLINICAL TRIAL: NCT06340243
Title: Risk Adapted Therapy of Hodgkin Lymphoma in Upper Egypt
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Enas Saad Hassan, principle investigator, Assiut University
Other Study IDs: HODGKIN
Record Dates: First submitted 2024-03-22; First posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2024-03

CONDITIONS: Pediatric Hodgkin Lymphoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radiotherapy — radiotherapy

SUMMARY:
determine if radiotherapy could be safely omitted for early hodgkin lymphoma responder patients without compromising outcome

DETAILED DESCRIPTION:
Hodgkin's lymphoma accounts for around 40% of all pediatric lymphomas and is the most prevalent cancer among adolescents and young adults. With combinations of chemotherapy and radiation, Hodgkin's lymphoma is roughly 80% curable, placing it among the most treatable cancers . Since the introduction of combination chemotherapy treatments 20 years ago, the prognosis for children with Hodgkin's lymphoma has improved. The treatment is mostly influenced by the stage of the disease at diagnosis, histology, existence of "B"-symptoms, and the presence of bulky disease. Nonetheless, 20% of patients do not achieve long-term remission, and around 20% experience treatment-related side effects such as secondary malignancies, infertility, cardiovascular disease, and organ malfunction following chemo-radiation .Studies of long-term therapy side effects were made possible by the significant number of survivors. The goal of therapy optimization protocols for pediatric patients with Hodgkin's lymphoma is to maintain excellent tumor control while limiting adverse effects and long-term consequences . It is critical to stratify patients based on reliable prognostic factors at presentation and according to the rapidity of response into low-risk (LR) patients who would benefit from less aggressive therapy, avoiding unnecessary toxic side effects, and high-risk (HR) patients who should be subjected to intensified therapy to reduce the rate of treatment failures and relapses .

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients younger than 18 years old with classical Hodgkin lymphoma

Exclusion Criteria:

* Patients aged more than 18 years old.
* Patients who died early at presentation before starting chemotherapy
* diagnosis of nodular lymphocytic predominant Hodgkin lymphoma
* previous chemotherapy or radiotherapy other (simultaneous) malignancies
* severe concomitant diseases (eg, immune deficiency syndrome); or known HIV positive.

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Infants and children around age of (1month to 18 years old) admitted with hodgkin lymphoma in a period of 2 years
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
assess the outcome of pediatric patients with HL treated with risk- and response-adjusted therapy | 2 years
  determine if radiotherapy could be safely omitted for early responder patients without compromising outcome, it can be assessed by decrease in lymph node volume ,Volumes are approximated as ellipsoids. If a, b, c denote the principal axes of the ellipsoid the volume is calculated as V= (a x b x c)/2